CLINICAL TRIAL: NCT05974865
Title: Amelioration of Literacy Deficits in Prenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HD050437; R01HD050437 (NIH)
Record Dates: First submitted 2014-07-22; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Prenatal Care; Health Literacy; Numeracy
Keywords: patient-physician communication; patient activation intervention; RIAS; health literacy; spoken literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Babies and Health Moms (Experimental): Healthy Babies and Healthy Moms was designed as a 20-minute communication skills-based computer program based on key social learning principles designed to empower women to more actively and productively use targetted skills to improve the medical dialogue of their prenatal visits.
  Interventions: Behavioral: Healthy Babies and Healthy Moms
- Baby Basics Prenatal Guide (Active Comparator): The Baby Basics Prenatal Guide, published by the What to Expect Foundation, was used in a face-to-face educational session with a study research assistant during which pregnancy related information was personalized by reviewing relevant sections of the Baby Basics prenatal guide.
  Interventions: Behavioral: Baby Basics Prenatal Guide

INTERVENTIONS:
Behavioral: Healthy Babies and Healthy Moms
  Arms: Healthy Babies and Health Moms
Behavioral: Baby Basics Prenatal Guide
  Arms: Baby Basics Prenatal Guide

SUMMARY:
The purpose of the study was to develop and evaluate a skill-based, computer intervention designed to facilitate effective prenatal visit communication for women with restricted literacy.

DETAILED DESCRIPTION:
The primary aim of the study is to develop and evaluate a skills-based, interactive computer intervention designed to enhance the communication skills of pregnant women with restricted literacy. To this end, a randomized trial compared a skill-based computer intervention to a facilitated review of pertinent print-based educational material on communication processes and its consequences. Intervention impact was evaluated through medical visit recordings and post-visit assessments by patients and clinicians. We hypothesized that women assigned to the skills-based, computer intervention would demonstrate greater use of targeted skills, be more actively engaged in the communication process, and experience more patient-centered visits than women assigned to the print-based intervention. We also hypothesized that computer use would result in greater visit satisfaction and closer patient and clinician alignment in their assessment of the patient's physical and emotional health status..

Study Design included 84 women seeing 19 obstetrical clinicians were randomized to use an interactive, skill-based, computer program or to a personalized review of a prenatal guide. Prenatal visits were recorded and coded using the Roter Interaction Analysis System (RIAS). Post-visit satisfaction and perceptions of physical and emotional health were reported. Analysis adjusted for the nesting of patients within physicians, gestation, literacy and visit length.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending study prenatal clinics with consenting clinicians. English speaking

Exclusion Criteria:

-

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2006-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
patient-centered communication | Baseline
  Audio recordings of the prenatal visits are coded using the Roter Interaction Analysis System (RIAS). The communication outcome measure is derived from this coding.

SECONDARY OUTCOMES:
depression as assessed by the Edinburgh Depression Scale | post medical visit up to 8 months
  The correlation between patient score on the The Edinburgh Depression Scale and the clinician's rating of signs of emotional state. The Edinburgh has 10 items items on a 4 point scale with score range 10-40. Higher scores indicating more symptoms of depression. Clinician completed a novel post visit assessment of the participant's emotional state asking to indicate signs of anxiety and depression observed during the recorded visit. 1 (no signs), 2 (some symptoms, but no illness), ), 3 (mild case), 4 (moderate case), 5 (severe case). Higher ratings indicated more significant anxiety and depression.

OTHER OUTCOMES:
patient satisfaction as assessed by a questionnaire developed by the study team | post medical visit up to 8 months
  Patient satisfaction with medical visit as assessed by a questionnaire developed by the study team. The measure consisted of 8 items on a 5-point scale ranging from poor (1) to excellent (5). Scale scores range from 8- 40.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Roter, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States